CLINICAL TRIAL: NCT00117689
Title: A Randomized, Controlled, Multi-Center Study of Thymoglobulin Induction Therapy With a Calcineurin Inhibitor Sparing Regimen in Liver Transplant Patients
Brief Title: Evaluation of Thymoglobulin Induction and Reduced Doses of Calcineurin Inhibitors on Liver Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Thymo102700103
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Liver Dysfunction; Rejection, Transplant; Transplantation, Liver
Keywords: Anti-T cell antibodies; Primary Liver Transplantation and Renal Dysfunction; Liver Transplant Rejection; Induction Therapy with reduction of Calcineurin inhibitors; Primary Liver Transplantation; Primary Transplant Rejection; Transplantation, Liver; Rejection, Transplant
MeSH Terms: conditions — Liver Diseases; Rejection, Psychology; Renal Insufficiency | interventions — thymoglobulin; Antilymphocyte Serum; Adrenal Cortex Hormones; Tacrolimus; Mycophenolic Acid

ARMS (2):
- 1 (Experimental): Standard (tacrolimus based standard therapy without induction)
  Interventions: Biological: Thymoglobulin; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- 2 Standard of Care (Active Comparator): Thymoglobulin with tacrolimus and corticosteroid sparing maintenance therapy
  Interventions: Drug: Corticosteroid; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Biological: Thymoglobulin — Antibody inductions with tacrolimus and corticosteroid sparing maintenance therapy
  Other Names: [Anti-thymocyte Globulin (rabbit)]
  Arms: 1
Drug: Corticosteroid — For a minimum of 3 months
  Arms: 2 Standard of Care
Drug: Tacrolimus — Between Day 3 the last dose of Thymoglobulin
Drug: Mycophenolate Mofetil — for at least 1 month posttransplant

SUMMARY:
This study involves the use of a drug called Thymoglobulin, which is approved in the US to treat kidney transplant rejection and in Canada to treat and prevent kidney transplant rejection. This study will evaluate the effect of Thymoglobulin induction therapy and reduced doses of calcineurin inhibitors on the incidence of liver rejection and will provide a basis for future evaluations of Thymoglobulin as an immunosuppressive agent to help decrease the incidence of liver transplant rejection. Subjects meeting all inclusion and exclusion criteria are eligible to participate in this study. Approximately 75 study subjects from up to 18 transplant centers in the United States and Canada will be enrolled in this 12-month study.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver transplant recipient with Model for End-Stage Liver Disease (MELD) criteria documentation
* Serum creatinine > 1.5mg/dL at the time of transplant, or based on the value used to calculate the most recent pre-operative MELD Score for liver allocation
* Ages greater than or equal to 18 years
* If female, must not be lactating; must have a negative serum beta-human chorionic gonadotropin (HCG) test within 7 days prior to Study Day 0 (Day of Transplant); and must agree to practice an acceptable and reliable form of contraception during the study
* Signed informed consent

Exclusion Criteria:

* Living donor or multiple organ transplants
* Prior solid organ or bone marrow transplant recipient
* Fulminant hepatic failure
* Status 1 transplants
* ABO incompatible transplants
* Transplants utilizing livers from non heart-beating donors
* Liver transplant candidates with > 6 weeks of analysis
* Donor with positive serology for hepatitis B surface antigen (HBsAg)
* Evidence of human immunodeficiency virus (HIV)
* Autoimmune hepatitis
* History of chronic steroid or immunosuppressant use in the 90 days prior to transplant, except for inhaled corticosteroids to treat asthma
* Recipient of investigational therapy within 90 days prior to transplant procedure
* Known contraindication to administration of rabbit anti-thymocyte globulin
* Acute viral illness
* History of malignancy within 5 years, with the exception of adequately treated localized squamous or basal cell carcinoma of the skin without evidence of recurrence, and/or hepatocellular carcinoma
* Illness other than primary liver disease (e.g. severe ischemic heart disease, left ventricular dysfunction, or pulmonary disease), which, in the opinion of the investigator, may significantly increase the risk of the transplantation procedure
* Current drug and alcohol abuse that, in the opinion of the investigator, puts subjects at risk for poor compliance (no drug test required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Freedom from biopsy-proven acute rejection (including humoral rejection) | 6 months

SECONDARY OUTCOMES:
Explore the impact of Thymoglobulin on kidney function after transplant | 6 months
Explore the impact of Thymoglobulin on the prevention of liver transplant rejection, transplanted liver loss, death, and safety of Thymoglobulin after transplant. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (16):
- United States (14):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - USC University Hospital, Los Angeles, California
  - University of California, San Fransisco Hospital, San Francisco, California
  - University of Colorado Hospital and Health Sciences Center, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Fairview University Medical Center, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, University Hospital, San Antonio, Texas
  - VCU Medical Center, Richmond, Virginia
- Canada (2):
  - Toronto University Hospital - UHN, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Thymoglobulin® — http://www.thymoglobulin.com/home/thymo_pdf_pi.pdf